CLINICAL TRIAL: NCT00529347
Title: The Effect of Positive End Expiratory Pressure (PEEP) on the Breathing Pattern During Neurally Adjusted Ventilatory Assist (NAVA)
Brief Title: Mechanical Ventilation Controlled by the Electrical Activity of the Patient's Diaphragm - Effects of Changes in Ventilator Parameters on Breathing Pattern
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Lukas Brander, MD, University Hospital Inselspital, Berne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SNF-3200B0-113478-1
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Mechanical Ventilation
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: neurally adjusted ventilatory assist (NAVA) — assessment of breathing pattern at various ventilator settings

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new concept of mechanical ventilation. NAVA delivers assist to spontaneous breathing based on the detection of the electrical activity of the diaphragm. We study the effect of changing ventilatory parameters on the patient's breathing pattern during NAVA.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation (tracheally intubated or tracheotomized)
* Presence of an arterial pressure line.
* Subject itself or its next of kin has given written informed consent

Exclusion Criteria:

* Patient is less than 18 years or more than 85 years of age
* The attending physician refuses to allow enrollment
* The patient refuses informed consent
* Next of kin is unavailable or refuses informed consent
* Pregnant or breast-feeding female. A pregnancy test will be performed in all female patients less than 60 years of age.
* Any contraindication to insertion/exchange a nasogastric tube, including (but not limited to): severe oropharyngeal malformation or bleeding; esophageal varices, tumor, infection, stenosis, or rupture
* Presence or suspicion of diaphragm injury
* Hemophilia or other severe bleeding disorder
* Presence or suspicion of a central nervous system (CNS) disorder, including (but not limited to): CNS infarction, bleeding, tumor, or infection
* History of heart and/or lung transplantation
* Any mechanical cardiac assist device (excluding intraaortic balloon pump)
* Any contraindication to reduce sedation or to stop neuromuscular blockage in order to allow spontaneous breathing
* The patient needs to be ventilated with a mode of mechanical ventilation that targets a predefined tidal volume or airway pressure as per attending physician
* Severe hemodynamic instability as per attending physician
* Planned or anticipated intervention within the study period necessitating either transfer out of the ICU or requiring prolonged interaction with the patient.
* A fraction of inspired oxygen (FiO2) of > 0.8
* The patient currently participates in another interventional clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in diaphragmatic Edi (area under the curve) during expiration | At each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Brander, MD, Principal Investigator — Department of Intensive Care Medicine, University Hospital, Bern, Switzerland
Locations (1):
- Department of Intensive Care Medicine, University Hospital - Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Derived] Passath C, Takala J, Tuchscherer D, Jakob SM, Sinderby C, Brander L. Physiologic response to changing positive end-expiratory pressure during neurally adjusted ventilatory assist in sedated, critically ill adults. Chest. 2010 Sep;138(3):578-87. doi: 10.1378/chest.10-0286. Epub 2010 Apr 30. PMID 20435654